CLINICAL TRIAL: NCT03182400
Title: Neurophysiological Study of Sensory and Cognitive Processes in Healthy Children and Adults
Acronym: PROSCEA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PHAO17-FBB/PROSCEA
Record Dates: First submitted 2017-05-23; First posted 2017-06-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteer (Experimental): Neurophysiological assessment Neuropsychological assessment
  Interventions: Behavioral: Neurophysiological assessment; Behavioral: Neuropsychological assessment

INTERVENTIONS:
Behavioral: Neurophysiological assessment — Assessment of cerebral electrical activity Assessment of ocular exploration Neurovegetative assessments
Behavioral: Neuropsychological assessment — sub-tests, scales, surveys, reaction time measurement

SUMMARY:
It is now widely accepted that autism is linked to a developmental disorder and cerebral function.

Our research team (UMR U930 INSERM, François-Rabelais University of Tours, whom Pr F Bonnet-Brilhault is responsible for team "Autism") hypothesizes that atypical sensory information processing, especially auditory and / or visual information, could underly the symptoms observed in autism. A better knowledge of the typical development of the sensory and cognitive processes must therefore make it possible in the long term to identify the abnormalities linked to the autism spectrum disorders (ASD).

Studies in healthy subjects are therefore necessary in order to identify neurophysiological indices of cerebral functioning and to study their evolution during normal development, making it possible in the future to compare with populations of subjects with ASD.

The investigators intend to study the development of all the cognitive processes involved in the processing of sensory and, in particular, auditory and visual information in humans: from low-level perception processes to higher-level cognitive processes (attention, emotion, language, prediction, ...). For this the investigators will use non-invasive neurophysiological explorations (EEG, eye tracking) as well as neuropsychological explorations (Questionnaires or spontaneous language recording).

A better understanding of the pathophysiological mechanisms underlying the symptoms observed in autism could ultimately lead to the development of new specific therapeutic strategies, particularly in the field of exchange and development therapy or cognitive remediation .

ELIGIBILITY:
Inclusion Criteria:

* Between 1 and 60 years-old
* Able to understand and apply instructions for a task
* Information of subject or legal representant
* Informed written consent of subject or legal representant
* Affiliation to the social security system

Exclusion Criteria:

* Abnormal corrected vision
* Abnormal audition
* Known personal neurological pathology
* Known personal psychiatric problems
* Identified difficulties for walking, language, or learning
* Exclusion period because of participation to another experimental protocol
* Adult with legal protection

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 450 (Estimated)
Dates: Start 2017-06-14 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
ERP amplitude (µV) | 1 hour
  analysis of ERP amplitude evoked during EEG recording

SECONDARY OUTCOMES:
Reaction times (ms) | 1 hour
  Reaction times collected during behavioral assessment
pupil size (mm) | 1 hour
  pupil size measurements acquired with the eye tracker

CONTACTS AND LOCATIONS:
Locations (1):
- Chru Tours, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided